CLINICAL TRIAL: NCT06727422
Title: A Phase 2b, Randomized, Double-Blind, Placebo- Controlled, Multicenter Study to Assess the Safety, Efficacy and Pharmacokinetics of RNIB21 in the Treatment of Patients With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: Efficacy of Rifaximin With NAC in IBS-D
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Pimentel, MD (Other)
Responsible Party: Sponsor-Investigator, Mark Pimentel, MD, staff physician II, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNIB21-201
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-12

CONDITIONS: IBS (Irritable Bowel Syndrome); IBS-D (Diarrhea-predominant)
Keywords: IBS-D
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- low dose for IBS-D (Experimental): RNIB21 containing rifaximin 66mg + NAC 560mg three times a day
  Interventions: Drug: rifaximin 66mg + N-acetylcysteine 560mg three times daily
- high dose for IBS-D (Experimental): RNIB21 containing rifaximin 132mg + NAC 560mg three times a day
  Interventions: Drug: RNIB21 containing rifaximin 132mg + N-acetylcysteine 560mg three times daily
- placebo (Placebo Comparator): placebo three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rifaximin 66mg + N-acetylcysteine 560mg three times daily — RNIB21 containing rifaximin 66mg + N-acetylcysteine 560mg three times daily
  Arms: low dose for IBS-D
Drug: RNIB21 containing rifaximin 132mg + N-acetylcysteine 560mg three times daily — RNIB21 containing rifaximin 132mg + N-acetylcysteine 560mg three times daily
  Arms: high dose for IBS-D
Drug: Placebo — placebo three times daily
  Arms: placebo

SUMMARY:
The purpose of this study is to examine the effectiveness of using a combination of a drug, rifaximin and a dietary supplement, N-acetyl-L-cysteine (NAC), to treat patients with irritable bowel syndrome with diarrhea (IBS-D). Rifaximin is one of the standard treatments for IBS-D and is FDA approved. While rifaximin is safe and effective for treating symptoms in patients with IBS-D, many patients find that their symptoms may not completely resolve, or may come back after a period of time.

This research study is designed to test the investigational use of a combination of rifaximin and NAC. The combination of rifaximin and NAC is not approved by the U.S. Food and Drug Administration (FDA) for the treatment of IBS-D, and the effects of taking both medications together are unknown. However, the two medications are approved for use separately, as detailed below.

Rifaximin is the only antibiotic approved by the FDA for the treatment of IBS-D. Rifaximin (at a dose of 550 mg by mouth three times daily for 14 days) is approved by the FDA for the treatment of IBS-D. Rifaximin (at a dose of 200 mg per mouth three times daily for 3 days) is FDA approved for the treatment of traveler's diarrhea. Rifaximin at a dose of 200 mg per mouth three times daily is not approved by the FDA for the treatment of IBS-D.

NAC is approved by the FDA to treat acetaminophen overdose (72-hour oral and 21-hour intravenous (IV) regimens), and for use in breaking up mucus in the lungs in patients with chronic obstructive pulmonary disease (COPD) and other lung conditions such as bronchitis. NAC is also available over-the-counter in 600 mg and 900 mg capsules as a dietary supplement, although over-the-counter use is not regulated by the FDA. This study will utilize the 600 mg dietary supplement capsules.

The Investigators want to know if using a combination of rifaximin and NAC will give better results in decreasing IBS-D symptoms than using rifaximin alone. As NAC is used to break up mucus in the lungs, and the Investigators want to see if this can also break up the mucus layer in the small intestine, and therefore potentially increase the effectiveness of rifaximin. The Investigators will be testing 2 doses to determine which dose is most effective.

participants are being asked to take part in this research study because participants were diagnosed with IBS-D.

DETAILED DESCRIPTION:
This is a phase 2b, multi-center, randomized, double-blind, placebocontrolled study of rifaximin in patients with IBS-D. Eligible patients will be randomized (1:1:1) to receive RNIB21 containing rifaximin 66mg + NAC 560mg TID; RNIB21 containing rifaximin 132mg + NAC 560mg TID; or placebo TID. The study will consist of the following phases: Screening Phase; Treatment Phase (Days 1 to 14) which includes the Randomization Visit (Day 1) and visits at Week 1 (Day 7 ± 2) and Week 2 (Day 14 ± 2); and a Follow-up Phase including an End of Study visit at Week 14 (Day 98 ± 3). REDCap, a web-based reporting system will be utilized to capture daily patient reported outcomes as regards abdominal pain and stool consistency. A subset of participating sites will be designated as Pharmacokinetics sites. In a blinded fashion 24 patients (8 from each treatment arm) will participate in PK sampling in order to establish a PK profile and PK parameters for both rifaximin and NAC. Serial blood samples will be collected following first dose and last dose to establish the PK profiles after a single dose, and multiple doses. The primary evaluation period (PEP) will be the 28 days following the completion of therapy. The primary outcome for the study will be adequate relief of IBS symptoms based on FDA guidance during this period, specifically: the proportion of patients who are responders to treatment in both IBS-related abdominal pain AND stool consistency during the 4-week PEP. A patient will be considered a weekly responder if there is adequate relief in their IBS-related symptoms, which is defined as a 30% or greater improvement from their baseline in the weekly average of worst abdominal pain in past 24 hours score AND at least 50% reduction in the number of days in a week with at least one stool that has a consistency of type 6 or 7 compared with their baseline. Responders have to meet both abdominal pain and stool consistency criteria for at least 2 of 4 weeks of the PEP. Abdominal pain will be self-reported on a daily basis using an 11-point (0-10) pain scale. Stool consistency will be self-reported daily by patients based on the Bristol Stool Scale. A smartphone app which captures stool image will be used as an seondary endpoint, and compared to the patients' self-reports of stool consistency recorded on the BSS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients ≥ 18 years of age
2. Diagnosed with IBS confirmed by the Rome IV criteria, with associated symptoms of diarrhea as noted below in 4(b).
3. Do not have adequate relief of IBS symptoms of abdominal pain, stool consistency or stool frequency
4. Have daily IBS symptom scores during screening as below:

   1. Weekly average score of worst daily abdominal pain >3.0 on a 0-10 point scale
   2. At least one stool with a consistency of Type 6 or 7 on the Bristol

Exclusion Criteria:

1. Present with the following symptoms of IBS with constipation:

   1. Less than 3 bowel movements a week,
   2. Hard or lumpy stools, and
   3. Excessive straining during a bowel movement.
2. History of inflammatory bowel disease, celiac disease, GI surgery (except cholecystectomy and/or appendectomy)
3. Evidence of active duodenal ulcer, gastric ulcer, diverticulitis, or active infectious gastroenteritis
4. Current diagnosis of asthma
5. Current user of NAC and/or rifaximin
6. Systemic antibiotic use in the last month
7. Not currently on a prokinetic drug
8. A significant medical condition including but not limited to hepatic, uncontrolled diabetes, renal, cardiovascular, pulmonary, uncontrolled thyroid disease. or psychiatric disease, which in the opinion of investigator precludes study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
stool consistency | 2 weeks
  A 50% reduction in the number of days per week with at least one stool consistency of Type 6 or 7 on the BSS compared to baseline, for at least 2 of the 4 weeks of the PEP
Abdominal pain | 2 weeks
  Abdominal pain will be self-reported on a daily basis using an 11-point (0-10) pain scale, where 10 represent the highest pain.;A 30% improvement compared to baseline on the weekly average score of worst daily abdominal pain for at least 2 of the 4 weeks of the primary evaluation period .

SECONDARY OUTCOMES:
overall response | up to 7 weeks of 14 weeks
  Overall response: Proportion of patients that achieve a weekly response during at least 50% of the weeks of treatment and follow up (i.e. 7 of 14 weeks
stool frequency | 2 weeks
  Stool frequency as number of bowel movements per day averaged on a weekly basis, versus baseline determined during the PEP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauritano EC, Gabrielli M, Lupascu A, Santoliquido A, Nucera G, Scarpellini E, Vincenti F, Cammarota G, Flore R, Pola P, Gasbarrini G, Gasbarrini A. Rifaximin dose-finding study for the treatment of small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2005 Jul 1;22(1):31-5. doi: 10.1111/j.1365-2036.2005.02516.x. PMID 15963077
- [Background] Scarpellini E, Gabrielli M, Lauritano CE, Lupascu A, Merra G, Cammarota G, Cazzato IA, Gasbarrini G, Gasbarrini A. High dosage rifaximin for the treatment of small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2007 Apr 1;25(7):781-6. doi: 10.1111/j.1365-2036.2007.03259.x. PMID 17373916
- [Background] O'Brien PC. Procedures for comparing samples with multiple endpoints. Biometrics. 1984 Dec;40(4):1079-87. PMID 6534410
- [Background] Pimentel M, Park S, Mirocha J, Kane SV, Kong Y. The effect of a nonabsorbed oral antibiotic (rifaximin) on the symptoms of the irritable bowel syndrome: a randomized trial. Ann Intern Med. 2006 Oct 17;145(8):557-63. doi: 10.7326/0003-4819-145-8-200610170-00004. PMID 17043337
- [Background] Sharara AI, Aoun E, Abdul-Baki H, Mounzer R, Sidani S, Elhajj I. A randomized double-blind placebo-controlled trial of rifaximin in patients with abdominal bloating and flatulence. Am J Gastroenterol. 2006 Feb;101(2):326-33. doi: 10.1111/j.1572-0241.2006.00458.x. PMID 16454838
- [Background] Trespi E, Ferrieri A. Intestinal bacterial overgrowth during chronic pancreatitis. Curr Med Res Opin. 1999;15(1):47-52. doi: 10.1185/03007999909115173. PMID 10216811
- [Background] Di Stefano M, Malservisi S, Veneto G, Ferrieri A, Corazza GR. Rifaximin versus chlortetracycline in the short-term treatment of small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2000 May;14(5):551-6. doi: 10.1046/j.1365-2036.2000.00751.x. PMID 10792117
- [Background] Corazza GR, Ventrucci M, Strocchi A, Sorge M, Pranzo L, Pezzilli R, Gasbarrini G. Treatment of small intestine bacterial overgrowth with rifaximin, a non-absorbable rifamycin. J Int Med Res. 1988 Jul-Aug;16(4):312-6. doi: 10.1177/030006058801600410. PMID 3169375
- [Background] Miglio F, Valpiani D, Rossellini SR, Ferrieri A. Rifaximin, a non-absorbable rifamycin, for the treatment of hepatic encephalopathy. A double-blind, randomised trial. Curr Med Res Opin. 1997;13(10):593-601. doi: 10.1185/03007999709113333. PMID 9327194
- [Background] Gillis JC, Brogden RN. Rifaximin. A review of its antibacterial activity, pharmacokinetic properties and therapeutic potential in conditions mediated by gastrointestinal bacteria. Drugs. 1995 Mar;49(3):467-84. doi: 10.2165/00003495-199549030-00009. PMID 7774516
- [Background] Attar A, Flourie B, Rambaud JC, Franchisseur C, Ruszniewski P, Bouhnik Y. Antibiotic efficacy in small intestinal bacterial overgrowth-related chronic diarrhea: a crossover, randomized trial. Gastroenterology. 1999 Oct;117(4):794-7. doi: 10.1016/s0016-5085(99)70336-7. PMID 10500060
- [Background] Nayak AK, Karnad DR, Abraham P, Mistry FP. Metronidazole relieves symptoms in irritable bowel syndrome: the confusion with so-called 'chronic amebiasis'. Indian J Gastroenterol. 1997 Oct;16(4):137-9. PMID 9357184
- [Background] Pimentel M, Chow EJ, Lin HC. Normalization of lactulose breath testing correlates with symptom improvement in irritable bowel syndrome. a double-blind, randomized, placebo-controlled study. Am J Gastroenterol. 2003 Feb;98(2):412-9. doi: 10.1111/j.1572-0241.2003.07234.x. PMID 12591062
- [Background] Drossman DA, McKee DC, Sandler RS, Mitchell CM, Cramer EM, Lowman BC, Burger AL. Psychosocial factors in the irritable bowel syndrome. A multivariate study of patients and nonpatients with irritable bowel syndrome. Gastroenterology. 1988 Sep;95(3):701-8. doi: 10.1016/s0016-5085(88)80017-9. PMID 3396817
- [Background] Agreus L, Svardsudd K, Nyren O, Tibblin G. Irritable bowel syndrome and dyspepsia in the general population: overlap and lack of stability over time. Gastroenterology. 1995 Sep;109(3):671-80. doi: 10.1016/0016-5085(95)90373-9. PMID 7657095
- [Background] Hungin AP, Whorwell PJ, Tack J, Mearin F. The prevalence, patterns and impact of irritable bowel syndrome: an international survey of 40,000 subjects. Aliment Pharmacol Ther. 2003 Mar 1;17(5):643-50. doi: 10.1046/j.1365-2036.2003.01456.x. PMID 12641512
- [Background] El-Serag HB. Impact of irritable bowel syndrome: prevalence and effect on health-related quality of life. Rev Gastroenterol Disord. 2003;3 Suppl 2:S3-11. PMID 12775997
- [Background] Gwee KA, Wee S, Wong ML, Png DJ. The prevalence, symptom characteristics, and impact of irritable bowel syndrome in an asian urban community. Am J Gastroenterol. 2004 May;99(5):924-31. doi: 10.1111/j.1572-0241.2004.04161.x. PMID 15128362
- [Background] Ruben H. A universally applicable dental prop. Br Dent J. 1968 Jun 4;124(11):525-6. No abstract available. PMID 5239910
- [Background] Bommelaer G, Poynard T, Le Pen C, Gaudin AF, Maurel F, Priol G, Amouretti M, Frexinos J, Ruszniewski P, El Hasnaoui A. Prevalence of irritable bowel syndrome (IBS) and variability of diagnostic criteria. Gastroenterol Clin Biol. 2004 Jun-Jul;28(6-7 Pt 1):554-61. doi: 10.1016/s0399-8320(04)95011-7. PMID 15243388
- [Background] Pimentel M, Chow EJ, Lin HC. Eradication of small intestinal bacterial overgrowth reduces symptoms of irritable bowel syndrome. Am J Gastroenterol. 2000 Dec;95(12):3503-6. doi: 10.1111/j.1572-0241.2000.03368.x. PMID 11151884
- See also: Read NW. Irritable Bowel Syndrome. In: Feldman J, Friedman LS, Sleisenger MH, eds. Sleisenger and Fordtran's Gastrointestinal and Liver Disease: Pathophysiology/Diagnosis/Management. 7th ed. Philadelphia, PA: Saunders; 2002: 1794-1806. — https://www.us.elsevierhealth.com/sleisenger-and-fordtrans-gastrointestinal-and-liver-disease-2-volume-set-9780323609623.html?srsltid=AfmBOopn8f9oC93B3DHlqQ4XZanoUyTPMubARrE7TOrzOXLt2uUQSD_R
- See also: Pimentel M. A New IBS Solution: Bacteria - The missing link in treating irritable bowel syndrome. Sherman Oaks, CA: Health Point Press; 2006. — https://books.google.com/books/about/A_New_IBS_Solution.html?id=0GJ6AAAACAAJ